CLINICAL TRIAL: NCT07218601
Title: Electronic Nose (E-nose) Technology to Assess Pathologic Response and Post- Treatment Progression for Non-small Cell Lung Cancer: a Phase II Study
Brief Title: Using E-Nose Technology to Track Treatment Response in People With Non-Small Cell Lung Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 25-124
Record Dates: First submitted 2025-10-16; First posted 2025-10-20 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: Non-Small Cell Lung Cancer
Keywords: E-Nose Technology; 25-124
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cohort 1 (stage II to IIIB NSCLC) (Experimental): 40 patients undergoing neoadjuvant treatment (stages II to IIIB) will undergo breath sampling (1) at baseline before any treatment, (2) 2 weeks after neoadjuvant therapy, (3) 2 weeks after surgery, (4) 6 months after surgery, and (5) every 6 months for the first 2 years. Blood sample collections will coincide with the breath collection schedule.
  Interventions: Diagnostic Test: Breath sample collection; Diagnostic Test: Research blood collection
- Cohort 2 (stage I NSCLC) (Experimental): 10 patients who are planned to undergo upfront surgery will undergo breath sampling (1) at baseline before upfront surgery, (2) 2 weeks after surgery, (3) 6 months after surgery, and (4) every 6 months for the first 2 years.
  Interventions: Diagnostic Test: Breath sample collection

INTERVENTIONS:
Diagnostic Test: Breath sample collection — Cohort 1: patients undergoing neoadjuvant treatment (stages II to IIIB) will undergo breath sampling (1) at baseline before any treatment, (2) 2 weeks after neoadjuvant therapy, (3) 2 weeks after surgery, (4) 6 months after surgery, and (5) every 6 months for the first 2 years.
  Cohort 2: patients who are planned to undergo upfront surgery will undergo breath sampling (1) at baseline before upfront surgery, (2) 2 weeks after surgery, (3) 6 months after surgery, and (4) every 6 months for the first 2 years.
Diagnostic Test: Research blood collection — Cohort 1: Blood sample collections will coincide with the breath collection schedule.
  Arms: Cohort 1 (stage II to IIIB NSCLC)

SUMMARY:
The researchers are doing this study to test the ability of a new technology called breathprinting, or electronic nose (E-Nose), to measure changes in certain chemicals in the breath before and after standard neoadjuvant therapy in people with NSCLC.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18
* Untreated clinical stage I NSCLC amenable to upfront surgery
* Untreated stage II to IIIB NSCLC amenable to neoadjuvant treatment followed by surgery
* ECOG Performance Status of ≤2 Of note, the E-nose is a completely noninvasive technology (only breath samples are collected). Therefore, this intervention would have no effects on a developing human fetus. There are therefore no requirements for the study population related to contraception or pregnancy testing.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-10-10 (Actual); Primary Completion 2027-10 (Estimated); Study Completion 2027-10 (Estimated)

PRIMARY OUTCOMES:
pathological response (Cohort 1: stages II to IIIB) | up to 2 years
  obtained using E-nose technology, all patients who have pre- and at least one post-neoadjuvant treatment E-nose testing performed will be considered evaluable for the primary endpoint of Major Pathologic Response (MPR). Patients with MPR confirmed on pathologic analysis will be considered to have had an MPR, whereas all other evaluable patients will be considered to have not had an MPR, in accordance with the intention-to-treat analysis.
progression (Cohort 1: stages II to IIIB) | up to 2 years
  Differences in VOC expression between time-point assessments will be calculated in terms of VOC percentage change from baseline to assess the magnitude of change among patients with and without progression, particularly at earlier time points. Here, progression is considered as a binary endpoint, where progression includes recurrence, disease progression, or death within 2 years.
progression (Cohort 2: Stage I) | up to 2 years
  Differences in VOC expression between time-point assessments will be calculated in terms of VOC percentage change from baseline to assess the magnitude of change among patients with and without progression, particularly at earlier time points. Here, progression is considered as a binary endpoint, where progression includes recurrence, disease progression, or death within 2 years.

CONTACTS AND LOCATIONS:
Overall Officials: Gaetano Rocco, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (7):
- United States (7):
  - Memorial Sloan Kettering Basking Ridge (All Protocol Activities), Basking Ridge, New Jersey
  - Memorial Sloan Kettering Monmouth (All Protocol Activities), Middletown, New Jersey
  - Memorial Sloan Kettering Bergen (All Protocol Activities), Montvale, New Jersey
  - Memorial Sloan Kettering Suffolk-Commack (All Protocol Activities), Commack, New York
  - Memorial Sloan Kettering Westchester (All Protocol Activities), Harrison, New York
  - Memorial Sloan Kettering Cancer Center (All Protocol Activities), New York, New York
  - Memorial Sloan Kettering Nassau (All Protocol Activities), Uniondale, New York

IPD SHARING:
Plan to Share IPD: Yes
Memorial Sloan Kettering Cancer Center supports the international committee of medical journal editors (ICMJE) and the ethical obligation of responsible sharing of data from clinical trials. The protocol summary, a statistical summary, and informed consent form will be made available on clinicaltrials.gov when required as a condition of Federal awards, other agreements supporting the research and/or as otherwise required. Requests for deidentified individual participant data can be made beginning 12 months after publication and for up to 36 months post publication. Deidentified individual participant data reported in the manuscript will be shared under the terms of a Data Use Agreement and may only be used for approved proposals. Requests may be made to: crdatashare@mskcc.org.

REFERENCES:
- See also: Memorial Sloan Kettering Center — https://www.mskcc.org/